CLINICAL TRIAL: NCT00837772
Title: Total Knee Replacement Using Standard Knee Cutting Guides vs Otismed MRI Generated Cutting Guide
Brief Title: Total Knee Replacement Study Using Standard Cutting Guide vs Otismed MRI Generated Cutting Guide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dossett01
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: Alignment
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Usual standard cutting guide for TKA (Total Knee Arthroscopy)
  Interventions: Device: Standard cutting guide for TKA
- Arm 2 (Experimental): Otismed MRI generated cutting guide for TKA
  Interventions: Device: Otismed MRI generated cutting guide for TKA

INTERVENTIONS:
Device: Standard cutting guide for TKA — Use of the usual cutting guide for surgical replacement of a diseased knee
  Arms: Arm 1
Device: Otismed MRI generated cutting guide for TKA — Use of the customized MRI generated cutting guide for surgical replacement of a diseased knee
  Other Names: Otismed
  Arms: Arm 2

SUMMARY:
Patients are referred to the VA orthopedic surgical clinic because of osteoarthritis and are requesting consideration for a total knee replacement. Those who qualify for the knee replacement are informed about the study. Those who consent to participate are randomly assigned to either the standard cutting guide or to the new method which is a MRI generated cutting guide called Otismed. All patients have an MRI so both groups will be unaware of which surgical technique is used. All patients receive the usual pre-op care and same type of replacement knee. Follow-up research visits are scheduled at 4 weeks, 3 and 6 months, and 1 and 2 years. Patients will be informed of which surgical technique they were randomized to at the conclusion of the study.

DETAILED DESCRIPTION:
Objective(s):

Primary:

Compare the surgical and clinical outcomes between patients receiving total knee replacement after random assignment to one of two groups:

1. surgical procedure with the standard knee cutting guide and
2. surgical procedure with the Otismed MRI generated cutting guide

Secondary:

Evaluate the cost benefit ratio related to the two different cutting guide uses.

Research Plan: All patients that are referred to orthopedics, are eligible for a total knee replacement for osteoarthritis and meet study criteria will be invited to participate. Patients will be randomly assigned to either the standard or the Otismed group. All patients will have a MRI of the knee. Patients and the research staff conducting measurements will be blinded to the type of cutting guide used for the surgery.

Methods: The study will be a randomized trial with the patient and data collector blinded to type of cutting guide used for the surgical procedure. The study will be conducted at one site and enrollment goal is 100 patients. Data collection will be done preoperatively and at 4 wks, 3 months, 6 months, one year and two year. Established instruments, the (Western Ontario and McMaster Universities Osteoarthritis Index) Womac and Oxford Knee Score, will be used. Measurements will be done to evaluate ROM (Range Of Motion) and assess post-op recovery. Surgical data and hospitalization data will be used for analysis of costs. Statistical analysis will be used for comparison of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All Veterans that are referred to orthopedics surgical clinic for a total knee replacement for osteoarthritis and meet study criteria will be invited to participate.

Exclusion Criteria:

* Patients who have undergone osteotomy, had previous healed tibia or femur fractures, previous joint replacement surgery or cannot have an MRI will be excluded.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2012-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Patient scores on Oxford, Womac, and Knee Society scores | 4 week, 3 mo. 6 mo. 1 yr. 2 yr.

SECONDARY OUTCOMES:
Leg alignment based on Long Leg CT scans | Post-op

CONTACTS AND LOCATIONS:
Overall Officials: Harold G. Dossett, MD MBA, Principal Investigator — Carl T. Hayden VA Medical Center
Locations (2):
- United States (2):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dossett HG, Estrada NA, Swartz GJ, LeFevre GW, Kwasman BG. A randomised controlled trial of kinematically and mechanically aligned total knee replacements: two-year clinical results. Bone Joint J. 2014 Jul;96-B(7):907-13. doi: 10.1302/0301-620X.96B7.32812. PMID 24986944
- [Derived] Dossett HG, Arthur JR, Makovicka JL, Mara KC, Bingham JS, Clarke HD, Spangehl MJ. A Randomized Controlled Trial of Kinematically and Mechanically Aligned Total Knee Arthroplasties: Long-Term Follow-Up. J Arthroplasty. 2023 Jun;38(6S):S209-S214. doi: 10.1016/j.arth.2023.03.065. Epub 2023 Mar 30. PMID 37003458